CLINICAL TRIAL: NCT02907749
Title: Effects of Spironolactone on Fibrosis Progression and Portal Pressure in Patients With Advanced Chronic Liver Disease
Brief Title: Spironolactone on Fibrosis Progrssion-Portal Hypertension(FP-PH)in Cirrhosis
Acronym: FP-PH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changqing Yang (Other)
Responsible Party: Sponsor-Investigator, Changqing Yang, MD, PhD, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Yang-20160905
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Spironolactone; Carvedilol; Combined Modality Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol (Active Comparator): Carvedilol starts at 6.25mg/d and increases to 12.5mg/d in next week as a maintainence dose
  Interventions: Drug: Spironolactone and carvedilol
- Spironolactone and carvedilol (Experimental): 1. Carvedilol starts at 6.25mg/d and increases to 12.5mg/d in next week as a maintainence dose
  2. Spironolactone is added after carvedilol being tolerated, which starts with 20mg/d and increases to 40mg/d as a maintainence dose
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Spironolactone and carvedilol — Patients are treated with carvedilol in combination with spironolactone.
  Other Names: Combination therapy
  Arms: Carvedilol
Drug: Carvedilol — Patients are treated with carvedilol only.
  Other Names: Single therapy
  Arms: Spironolactone and carvedilol

SUMMARY:
The aim of this study is to investigate the effects of spironolactone on liver fibrosis progression and portal pressure gradient in patients with advanced chronic liver disease. Eligible cirrhosis patients were 2:1 randomized to either combination (carvedilol and spironolactone) or single (carvedilol) therapy group. Changes in virtual portal pressure gradient (vPPG) of portal trunk (calculated based on reconstructed 3D model and measured blood flow velocity), liver stiffness measurement (Fibroscan) and serum markers of liver fibrogenesis were documented at baseline and six months later.

ELIGIBILITY:
Inclusion Criteria:

-Proven cirrhosis based on histology or unequivocal clinical, sonographic and laboratory findings

Exclusion Criteria:

* Treatment with β-blockers or diuretics in the last 3 months
* Severe cardiopulmonary or renal insufficiency
* Chronic alcohol abuse
* Can't tolerate side effects of oral carvedilol or spironolactone
* History of variceal bleeding
* Malignancy
* Portal vein thrombosis
* History of partial splenic embolization or splenectomy
* Moderate or tense ascites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Virtual portal pressure gradient(vPPG) | 6 months
  Calculated based on reconstructed 3D portal trunk using anatomical information extracted from CT angiography and blood flow velocity measured by Doppler ultrasound

SECONDARY OUTCOMES:
Liver stiffness measurement (LSM) | 6 months
  Detected using FibroScan
Occurence of portal hypertension-related complications | 6 months
  variceal bleeding, ascites, hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, M.D., Study Director — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Tongji University, Shanghai, Shanghai Municipality, China